CLINICAL TRIAL: NCT02923063
Title: A Randomized, Controlled Trial of Personalized, Home-based Exercise Training on Muscle Mitochondrial Function and Metabolism
Brief Title: Exercise Study Testing Enhanced Energetics of Mitochondria Video Integrated Delivery of Activity Training in CKD
Acronym: ESTEEM-VIDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1343904
Record Dates: First submitted 2016-09-29; First posted 2016-10-04 (Estimated); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Moderate-severe Chronic Kidney Disease Not Treated With Dialysis; Diabetic Kidney Disease, HgbA1c Less Than 8.5
Keywords: Chronic Kidney Disease; Mitochondrial Metabolism; Physical Performance; Exercise Intolerance; Muscle Fatigue
MeSH Terms: conditions — Diabetic Nephropathies; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Aerobic and Resistance Exercise (Experimental): Exercise will be supervised by exercise trainers 3 days per week for 12 weeks via videoconferencing. Each session will start at 30 minutes in duration and include either high-intensity interval targeting a relative perceived exertion (RPE) of greater than 14 (on a scale of 6-20) or strength training (RPE 12-14) or power walking (RPE 12-14). Each 1 week of supervised sessions will alternate with 1 week of self-directed sessions with mid-week trainer check-in.
  Interventions: Behavioral: Combined Aerobic and Resistance Exercise via videoconferencing
- Usual Care (No Intervention): The control group will receive a one-time counseling session on appropriate dietary and physical activity recommendations. They will receive a "Go4Life Workout to go" sample exercise routing created by the national institutes on aging (NIA).

INTERVENTIONS:
Behavioral: Combined Aerobic and Resistance Exercise via videoconferencing — Combined aerobic and resistance exercise session thrice weekly for 12 weeks
  Arms: Combined Aerobic and Resistance Exercise

SUMMARY:
Skeletal muscle dysfunction (sarcopenia) is an under-recognized target organ complication of CKD with substantial adverse clinical consequences of disability, hospitalization, and death. Sarcopenia in this proposal is defined by impaired metabolism and physical function associated with decreased skeletal muscle mass or function. Skeletal muscle tissue relies on mitochondria to efficiently utilize oxygen to generate ATP. Impaired mitochondrial energetics is a central mechanism of sarcopenia in CKD. The investigators propose a series of studies designed to shed light on the pathophysiology of sarcopenia in persons with CKD not treated with dialysis. Investigators will conduct a randomized-controlled intervention trial of combined resistance training and aerobic exercise vs. health education to assess changes in skeletal muscle mitochondrial function, metabolism and physical function. Investigators hypothesize that exercise improves mitochondrial function and physical function in persons with CKD. If successful, these experiments will identify novel pathophysiologic mechanisms for CKD-associated sarcopenia. The proposed study will provide useful insight into benefits associated with exercise among patients with CKD and investigate mechanisms associated with improved metabolism, muscle function and physical function in population.

DETAILED DESCRIPTION:
Sarcopenia is a common complication of chronic kidney disease. Sarcopenia is defined by decreased muscle mass or function and is central to the frailty phenotype that is associated disability, hospitalization, and death. Sarcopenia is a common and devastating complication of chronic kidney disease (CKD). The investigators and others have demonstrated a high prevalence of physical frailty among CKD patients not treated with dialysis. Furthermore the investigators have demonstrated greater than 30% impairment in lower extremity physical performance measures in persons with CKD compared with predicted values. The aging demographic among CKD patients will result in a substantial U.S. public health burden attributable to sarcopenia. In the year 2000, direct healthcare costs attributable to sarcopenia in the U.S. were18.5 billion.

Sarcopenia is associated with adverse health-related outcomes. Sarcopenia in older adults is consistently linked with decreased physical functioning, disability, falls, hospitalization, and mortality. Impaired lower extremity physical performance, as measured by objective testing, is associated with all-cause mortality in CKD patients not treated with dialysis and that these associations are stronger in magnitude than those for traditional risk factors. Skeletal muscle is major site of peripheral glucose utilization ameliorating oxidative stress and endothelial injury associated with acute post-prandial hyperglycemia. Through these mechanisms sarcopenia may contribute to metabolic disturbances of insulin resistance, oxidative stress, and endothelial dysfunction leading to cardiovascular disease.

Mitochondrial dysfunction is central to skeletal muscle dysfunction. Skeletal muscle mitochondria are necessary for the efficient generation of energy (ATP) from oxygen and normal lipid metabolism. Under normal conditions, muscle efficiently utilizes the majority of supplied oxygen such that only 0.2% of mitochondrial oxygen is shuttled into reactive oxidative species (ROS). Under pathologic situations there is uncoupling of oxygen consumption and ATP generation resulting in increased oxygen consumption and decreased ATP production in a process leading to increased ROS and oxidative stress. Uncoupling of oxygen and ATP generation directly affects skeletal muscle function. Decreased efficiency of ATP generation has been linked to decreased muscle strength and more recently associated with decreased gait speed in older adults.

Magnetic resonance spectroscopy and optical spectroscopy (MRS/OS) provide novel, non-invasive and real-time insight into human skeletal muscle mitochondrial function. MRS/OS is a novel technique that measures maximal mitochondrial ATP production in-vivo following acute bouts of ischemia induced by exercise using phosphorous MRS (31P MRS). The rate of recovery of phosphocreatinine after cessation of exercise is used to characterize the rate of aerobic mitochondrial ATP resynthesis above that of basal anaerobic glycolytic ATP production. By combining this technique with optical spectroscopy post-exercise measuring the transport of oxygen from hemoglobin to myoglobin within the muscle the investigators are able to accurately determine the ratio of coupling efficiency between of ATP generation per unit of oxygen consumption. Skeletal muscle mitochondrial dysfunction measured by ATP generating capacity and coupling efficiency has been associated with processes of aging and insulin resistance. Furthermore studies in healthy subjects have shown that muscle performance and fatigue are linked to the ability to resynthesize ATP rather than lactate concentration.

Preliminary MRS/OS findings suggest profoundly altered mitochondrial function in CKD patients. Previous experimental studies suggest that uremia in dialysis patients affects skeletal muscle structure and mitochondrial function. Oxidative damage is highly prevalent in CKD, evidenced by increased biomarkers of oxidative stress and changes in glutathione, an important antioxidant. Prior small studies in non-diabetic CKD patients suggest impairment of ex-vivo mitochondrial function by reductions in mitochondrial enzyme activity. Based on these findings investigators used novel, non-invasive, functional MRS/OS assay to characterize in-vivo mitochondrial function. Preliminary findings in non-diabetic CKD patients indicate markedly reduced ATP to oxygen ratio compared to controls. This finding suggests altered mitochondrial energetics as a candidate central mechanism linking metabolic derangements and impaired physical function in CKD, and motivate the hypothesis that mitochondrial dysfunction is associated with oxidative stress, insulin resistance and impaired physical functioning in CKD.

Exercise may ameliorate mitochondrial dysfunction, insulin resistance and physical functioning in CKD. Studies of exercise in non-CKD patients with diabetes and insulin resistance have demonstrated exercise-induced improvements in mitochondrial biogenesis linked to improved insulin sensitivity as well as decreased mitochondrial oxidative stress. Animal studies suggest that exercise stimulates autophagy resulting in removal of defective and inefficient mitochondrial leading to a healthy mitochondrial network and improved insulin sensitivity.The primary goal of this study is to investigate the impact of combined resistance and aerobic exercise on skeletal muscle dysfunction. Given the investigator's preliminary data demonstrating strong association of sarcopenia and mortality in CKD, effective interventions that can impact physical function are urgently needed to improve patient health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-severe CKD determined by estimated glomerular filtration rate (eGFR) <60ml/min per 1.73m2
* No history chronic treatment with dialysis.
* Age 30 years old to 75 years
* Sedentary defined as self-reporting no more than 1 day per week of regular (structured) endurance exercise (EE) [e.g., brisk walking, jogging/running, cycling, elliptical, or swimming activity that results in feelings of increased heart rate or rapid breathing (EE), and/or sweating] or resistance exercise (RE) (resulting in muscular fatigue) lasting no more than 60 minutes in the past year.

  * Persons bicycling as a mode of transportation to/from work > 1 day/week etc. are not considered sedentary
  * Leisure walkers are included unless they meet the heart rate, breathing and sweating criteria noted above
  * Persons adherent to both 1 day/week of RE and 1 day/week of EE are excluded

Exclusion Criteria:

* Current or previous transplantation
* Current pregnancy (all females of child-bearing potential will have a pregnancy test)
* Wheelchair dependence or other disability that precludes physical exercise
* Oxygen dependent Chronic obstructive pulmonary disease (COPD)
* Shortness of breath after walking <100 steps on flat surface
* Weight >300 pounds
* HIV infection or hepatitis viral infection
* Decompensated cirrhosis
* Active malignant cancer other than non-melanomatous skin cancer
* Drugs that alter mitochondrial function:

  * muscle relaxants (methocarbamol, baclofen, tizanidine, carisoprodol, cyclobenzaprine)
  * oral steroids (Equivalent of 10mg or more of prednisone daily)
  * anti-viral medications (tenofovir, zalcitabine, didanosine, stavudine, lamivudine, zidovudine, abacavir, adefovir, interferon, ribavirin, efavirenz, dasabuvir, ombitasvir)
  * oral calcineurin inhibitors (Tacrolimus, Cyclosporine)
  * Antiepileptic drugs (Phenytoin, phenobarbital, carbamazepine, valproic acid, oxcarbazepine, ethosuximide, zonisamide, topiramate, and vigabatrin)
  * Antipsychotics (haloperidol, thioridazine, risperidone, quetiapine, clozapine, olanzapine and aripiprazole)
* Drugs- anticoagulants or antiplatelets

  * Anticoagulants, any 1 (coumadin, rivaroxaban, apixaban, dabigatran, edoxaban)
  * Antiplatelets, any 2 (aspirin, cilostazol, clopidogrel, dipyridamole, prasugrel, ticagrelor, ticlopidine, vorapaxar)
* Implants that prohibit MRI measurements or trauma involving metal fragments
* Pacemaker
* History of clotting disorder (Deep venous thrombosis, pulmonary embolism) or bleeding disorder.
* History of sever heart disease/disorders: coronary artery bypass graft (CABG) surgery, atrial fibrillation
* Vascular stent: bare metal or any recently placed (within 6 months)
* Current substance abuse
* Institutionalization
* Current participation in an interventional trial
* Inability to provide informed consent without a proxy respondent
* Non-English speaking
* Any condition which in the judgement of the clinical investigator places the participant at risk from participation in the study.

Additional Criteria:

* On chronic dialysis
* Expectation to start dialysis within 6 months.
* High dose antioxidants (Vitamine C, Vitamin E)
* Baseline systolic blood pressure >170 or diastolic blood pressure >100
* Uncontrolled diabetes with a HgbA1c >8.5
* Active uncontrolled thyroid disease
* Anemia (Hgb <9 g/dL)
* Current substance abuse (i.e. amphetamine abuse)
* Chronic opioid use (i.e. for chronic pain)
* Chronic use of immunosuppressants
* Active coronary ischemia detected by ECG on cycle ergometry VO2max testing. These individuals will be promptly referred to their primary care provider by the PI.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Mitochondrial phosphorylation capacity (ATPmax) by in-vivo 31P MRS | 12 weeks
  leg muscles
Quadriceps muscle work efficiency | 12 weeks
  Work efficiency calculated by cycler ergometry VO2

SECONDARY OUTCOMES:
Change in physical performance | 12 weeks
  6 minute walking distance (meters)
Change in Systemic oxidative stress (markers of arachidonic acid peroxidation) | 12 weeks
  Plasma isofurans (pg/min)
Change in aerobic capacity (VO2max) (ml/kg/min) | 12 weeks
Monocyte bioenergetics | 12 weeks
  Reserve Capacity (pmole/min/mcg protein)
Total work | 12 weeks
  Total work performed on cycle ergometer (kilojoules)
Muscle mitochondrial reactive oxygen species production from muscle tissue. | 12 weeks
  ratio of hydrogen peroxide (H2O2) production (pmol/min/mg tissue) to oxygen consumption (pmol/min/mg protein)
Muscle mitochondrial oxidative phosphorylation capacity. | 12 weeks
  maximum oxygen consumption production (pmol O2/min/mg tissue) to oxygen consumption (pmol/min/mg protein)
Self-reported fatigue (NIH PROMIS Fatigue) | 12 weeks
  self reported fatigue
Self-reported physical function (PROMIS mobility) | 12 weeks
  self reported difficulty with mobility
MoCA test (cognitive testing) | 12 weeks
  self-reported cognitive testing
Connor-Davidson Resilience Scale 25 (CD-RISC-25) | 12 weeks
  self-reported cognitive testing (depression)
Health Questionnaire | 12 weeks
  self-reported personal health history
FACIT fatigue scale (Version 4) | 12 weeks
  self-reported fatigue scale
Physical Activity Questionnaire (HAP) | 12 weeks
  self reported activity
Lubben Social Network Scale | 12 weeks
  self-reported social engagement questionnaire
Pittsburgh Fatigability Scale | 12 weeks
  self-reported fatigability
Self-Efficacy for Managing Chronic Conditions (PROMIS Bank) | 12 weeks
  self-reported Managing Symptoms, Managing Emotions, Managing Medications and Treatment, Managing Social Interactions, Managing Daily Activities, Cognitive Function, and Profile
Kidney Disease and Quality of Life (KDQOL-SF™ 1.3) | 12 weeks
  self-reported kidney health
Perceived Stress (NIH) | 12 weeks
  self reported perceived stress

OTHER OUTCOMES:
Walking economy during 6 minute walk | 12 weeks
  Assessement of energetic cost of walking during a submaximal 6 minute walk test using COSMED

CONTACTS AND LOCATIONS:
Overall Officials: Baback Roshanravan, MD MS MSPH, Principal Investigator — UC Davis; Javier Lopez, MD, Principal Investigator — UC Davis Department of Medicine/Division of Cardiology
Locations (1):
- UC Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/exercise-and-energy-production-in-chronic-kidney-disease-study-671748/